CLINICAL TRIAL: NCT03086226
Title: A Randomized, Double Blind Phase II Proof-of-Concept Superiority Trial of Fosravuconazole 200 mg or 300 mg Weekly Dose Versus Itraconazole 400 mg Daily, All Three Arms in Combination With Surgery, in Patients With Eumycetoma in Sudan
Brief Title: Proof-of-Concept Superiority Trial of Fosravuconazole Versus Itraconazole for Eumycetoma in Sudan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DNDi-FOSR-04-MYC
Record Dates: First submitted 2017-01-25; First posted 2017-03-22 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Mycetoma
Keywords: Mycetoma Fosravuconazole Itraconazole Surgery Sudan
MeSH Terms: conditions — Mycetoma | interventions — fosravuconazole L-lysine ethanolate; Itraconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fosravuconazole 300 mg (Experimental): Given throughout the study for 12 months as the experimental arm.
  Both experimental arms will be evaluated at 3 months. At this time-point, one of the study arms will be dropped according to the drop-the-loser design, based on efficacy or toxicity.
  Interventions: Drug: Fosravuconazole
- Fosravuconazole 200 mg weekly (Experimental): Given throughout the study for 12 months as the experimental arm.
  Both experimental arms will be evaluated at 3 months. At this time-point, one of the study arms will be dropped according to the drop-the-loser design, based on efficacy or toxicity.
  Interventions: Drug: Fosravuconazole
- Itraconazole 400mg daily (Active Comparator): Given throughout the study for 12 months as the comparator arm.
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: Fosravuconazole — Fosravuconazole will be given in two arms either as 300mg or 200mg. The drop-the loser design adaptive clinical trial design will allow two stages of the trial separated by a data based decision. In the first stage a decision will be taken on which arm to drop either the Fosravuconazole 200 or the Fosravuconazole 300 arm. The best treatment will be compared against the standard of care, itraconazole. At the end the focus will be comparing the best treatment against standard of care.
  Other Names: E1224
  Arms: Fosravuconazole 200 mg weekly; Fosravuconazole 300 mg
Drug: Itraconazole — This will be the active comparator
  Other Names: Sporanox
  Arms: Itraconazole 400mg daily

SUMMARY:
This study is a single-center, comparative, randomized, double-blind, parallel-group, active-controlled, clinical superiority trial of Fosravuconazole versus Itraconazole combined with surgery in subjects with eumycetoma in Sudan.

There will be three arms in this study: The first arm will be Fosravuconazole 300 mg weekly, the second arm will have Fosravuconazole 200 mg weekly and the control arm is the standard treatment using itraconazole 400mg daily.

At 3 months time-point, interim analysis will be done and one of the study arms will be dropped according to the drop-the-loser design, based on efficacy or toxicity.

DETAILED DESCRIPTION:
Eumycetoma is a fungal disease caused by Madurella mycetomatis. The disease is chronic, granulomatous and inflammatory. It usually involves subcutaneous tissues and leads to masses and sinuses from which fungal grains are discharged. It is most probably introduced post trauma e.g. thorn prick. It is associated with major morbidity and can be disabling, disfiguring and highly stigmatizing. In advanced cases it may be fatal. Eumycetoma is most prevalent in what is known as mycetoma belt.

Current treatment modalities for eumycetoma are disappointing. The response is characterized by low cure rates, high amputation rates, high up drop out from follow up and high recurrence rates. The available drugs for the treatment of eumycetoma are expensive, potentially toxic and require a long treatment period up to 12 months. By that time the mass is well encapsulated and is removed surgically. Despite prolonged medical treatment, the causative organisms are commonly found to still be viable and can be cultured from the surgical specimen.

The objectives of this study are to determine the comparative efficacy, safety, and tolerability of Fosravuconazole versus itraconazole as first-line treatment for subjects with eumycetoma caused by Madurella mycetomatis. The primary end-point will be complete cure after 12 months treatment as evidenced by clinical assessment showing absence of mycetoma mass with closure of sinuses and absent discharge, normal ultrasonic examination of the lesion, or the presence of fibrosis only associated with a negative fungal culture from a surgical biopsy from the former mycetoma site. The secondary endpoints are the outcome at 3-month's time point based on the same criteria as 12 month and/or treatment-related adverse events at the 3- and 12-month visits. The study will also monitor plasma drug levels of ravuconazole and itraconazole that will be included in a logistic model with other clinical and laboratory parameters to predict outcome. In addition, immunological studies will be done to describe the developing or changing immune responses during treatment. Lastly, all strains collected will be cultured and typed and with assessment of antifungal resistance.

This study is a single-center, comparative, randomized, double-blind, parallel-group, active-controlled, clinical superiority trial in subjects with eumycetoma requiring surgery. There will be three arms this study: The first arm will have Fosravuconazole 300 mg weekly and the second arm will have Fosravuconazole 200 mg weekly. Both arms will be evaluated at 3 months. At this time-point, one of the study arms will be dropped according to the drop-the-loser design, based on efficacy or toxicity. The control arm is the standard treatment using itraconazole 400mg daily. Patients will receive treatment for one year. An interim analysis is planned after data has been accumulated for sample size of 28 for 3 months end point.

This study will be done at the Mycetoma Research Centre, Sudan when ethics and regulatory approvals are received. The study plans to recruit 138 subjects by the end of the trial. The main inclusion criteria are subjects who provide consent, aged 18 years or more with primary moderate eumycetoma (size 2-10 cm) caused by Polymerase Chain Reaction (PCR) confirmed Madurella mycetomatis. Females in the child bearing age will require stringent contraception. The main exclusion criteria are eumycetoma > 10 cm, previous treatment, significant concomitant illness that preclude evaluation and treatments or conditions treated with drugs that are known to interact with the azoles.

The study is expected to new safer and more efficacious eumycetoma treatment.

ELIGIBILITY:
Inclusion Criteria

1. Participants with eumycetoma caused by M. mycetomatis confirmed by PCR.
2. Participants with eumycetoma requiring surgery.
3. Eumycetoma lesion ≥ 2 cm and < 16 cm in diameter. Note: A lesion was defined as either one single lesion on one anatomical area or multiple lesions on one anatomical area provided that the total affected area remained within the given limits.
4. Age ≥ 15 years.
5. Able to comply with protocol procedures and available for follow-up.
6. Written informed consent from the participant. If the participant was < 18 years old, there had to be a signed consent from a parent or legal guardian AND a written assent signed by the participant.
7. Female specific inclusion criteria:

   1. Negative pregnancy test.
   2. If women of childbearing potential (WOCBP), to use adequate contraception during the trial period until 2 months after completion of trial treatment.

Exclusion Criteria

1. Previous surgical or medical treatment for eumycetoma which included any previous antifungal treatment.
2. Presence of loco-regional lymphatic extension, osteomyelitis, other bone involvement based on radiology or any pre- or co-existing condition that could have precluded evaluation of the eumycetoma. Note: The presence of bone involvement would need a different treatment with a longer duration.
3. Pregnancy or lactation at screening, or intent to have become pregnant.
4. Concomitant or severe diseases that could have compromised the participant follow-up or evaluation (e.g., psychiatric condition, chronic hepatitis, neutropenia, human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS), diabetes mellitus or adrenocortical insufficiency).
5. Severe malnutrition as defined by a body mass index (BMI) < 16 kg/m2.
6. Contraindication to use itraconazole, including congestive heart failure, ventricular dysfunction, ventricular arrhythmia and negative inotropic state; Note: for a comprehensive list of contraindications and contraindicated concomitant medication refer to the package insert for itraconazole (Sporanox®);
7. Contraindication to the use of fosravuconazole;
8. Pre-existing liver disease, transaminase levels > 2x the laboratory's upper limit of normal (ULN) or elevated levels of alkaline phosphatase (ALP) or bilirubin.
9. Was receiving or likely to have required drugs that were either a substrate for cytochrome P450 family 3 subfamily A member 4 (CYP3A4) and/or metabolised by CYP3A4 (cisapride, oral midazolam, nisoldipine, felodipine, pimozide, quinidine, dofetilide, triazolam, methodone and levacetylmethadol [levomethadyl] were contraindicated);
10. Fridericia's corrected QT interval (QTcF) > 450 msec on any ECG known about or taken prior to trial entry.
11. Familial short QT syndrome or corrected QT interval (QTc) prolongation.
12. History of hypersensitivity to any azole antifungal drug.
13. Participation in other CTs within a 6-month period.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with complete cure at the End-of-Treatment | 12 months
  Complete cure at the End-of-Treatment (EOT; 52-week time point) in the Modified Intention to Treat (mITT) population.
  Complete cure of mycetoma is defined as
  1. negative fungal culture from a surgical biopsy from the former mycetoma site AND
  2. clinical cure (no clinical evidence of mycetoma mass, sinus tract, or discharge) AND
  3. normal lesion site or only fibrosis on sonogram

SECONDARY OUTCOMES:
Proportion of patients with complete cure of the Mycetoma at the end of the study | 15 months
  Complete cure of the mycetoma at the End Of Study (EOS; 15 months) visits Complete cure of mycetoma is defined as
  1. negative fungal culture from a surgical biopsy from the former mycetoma site AND
  2. clinical cure (no clinical evidence of mycetoma mass, sinus tract, or discharge) AND
  3. normal lesion site or only fibrosis on sonogram
Proportion of patients with mycological eradication of Mycetoma | 12 months
  Mycological eradication of the etiologic fungal pathogen from the mycetoma biopsy at the EOT visit (52-week time point). Mycological eradication is defined as negative Mycetoma culture biopsy.
Proportion of patients considered to have effective treatment at the End of Treament | 12 months
  Effective treatment (combination of mycological eradication AND clinical improvement in the mycetoma lesion) at EOT (52-week time point) visit in the mITT and Clinically Evaluable (CE) Populations.
  Mycetoma clinical improvement is defined by reduction in mycetoma mass size. Mycological eradication is defined as negative Mycetoma culture biopsy.
Proportion of patients considered to have effective treatment at the End of Study | 12 months
  Effective treatment (combination of mycological eradication AND clinical improvement in the mycetoma lesion) at EOS (15 months) visit in the mITT and Clinically Evaluable (CE) Populations.
  Mycetoma clinical improvement is defined by reduction in mycetoma mass size. Mycological eradication is defined as negative Mycetoma culture biopsy.
Propoprtion of patients with complete mycetoma cure by fungus genus at End of Treatment | 12 months
  Complete cure, effective treatment, and overall improvement categorized by etiologic fungal genus and species at EOT (52-week time point) visits in the mITT and CE populations
Propoprtion of patients with complete mycetoma cure by fungus genus at End of Study | 15 months
  Complete cure, effective treatment, and overall improvement categorized by etiologic fungal genus and species at EOS (15 months) visits in the mITT and CE populations
Immunological changes | 15 months
  Immunological parameters indicating a switch from a Th2 to a Th1 response. This includes measurement of cytokines, immunoglobulins and cells
Time to complete cure | 15 months
  The time to onset of cure will be calculate for each subject
Time to effective treatment | 15 months
  The time to effective treatment will be calculate for each subject (combination of mycological eradication and clinical improvement in the mycetoma lesion).
Time to failure | 15 months
  The time to relapse will be calculate for each subject
The proportion of subjects experiencing at least one Adverse Event | 15 months
  The safety consists the description of each serious adverse event and adverse event (preferred term) per treatment group and classified by system organ. ECG and Laboratory abnormalities will be considered as Adverse Events.
The frequency of the Adverse Events and Serious Adverse Events that lead to treatment discontinuation. | 15 months
  The safety consists the description of each serious adverse event and adverse event (preferred term) per treatment group and classified by system organ. ECG and Laboratory abnormalities will be considered as Adverse Events.
Severity of the Adverse Events and Serious Adverse Events that lead to treatment discontinuation. | 15 months
  The safety consists the description of each serious adverse event and adverse event (preferred term) per treatment group and classified by system organ. ECG and Laboratory abnormalities will be considered as Adverse Events.
CMax | 15 months
  Derived exposure parameters of ravuconazole and itraconazolecalculated from the final PK model using individual posterior estimates of the PK parameters and from dosing history.
AUC at steady-state (AUCss) | 15 months
  Derived exposure parameters of ravuconazole and itraconazolecalculated from the final PK model using individual posterior estimates of the PK parameters and from dosing history.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Fahal, Prof, Principal Investigator — Mycetoma Research Centre, Soba University, Khartoum, Sudan
Locations (1):
- Mycetoma Research Centre, Khartoum, Sudan

IPD SHARING:
Plan to Share IPD: Yes
Through Drugs for Neglected Diseases Initiative (DNDi) and open data sharing platforms. The data may be obtained by sending a request to DNDi
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 24 months of last subject last visit
Access Criteria: Data Requestors will enter into an appropriate agreement or terms of use and will adhere to contractual obligations
URL: http://dndi.org

REFERENCES:
- [Derived] Chu WY, Fahal AH, Ahmed ES, Bakhiet SM, Bakhiet OE, Fahal LA, Mohamed AA, Mohamedelamin ESW, Bahar MEN, Attalla HY, Siddig EE, Mhmoud NA, Musa AM, Oyieko P, Egondi T, Bruggemann RJ, Hata K, Strub-Wourgaft N, Alves F, Nyaoke BA, Zijlstra EE, Dorlo TPC. Pharmacokinetics and Pharmacodynamics of Fosravuconazole, Itraconazole, and Hydroxyitraconazole in Sudanese Patients With Eumycetoma. J Infect Dis. 2025 Sep 15;232(3):e518-e528. doi: 10.1093/infdis/jiaf279. PMID 40433693
- [Derived] Fahal AH, Ahmed ES, Bakhiet SM, Bakhiet OE, Fahal LA, Mohamed AA, Mohamedelamin ESW, Bahar MEN, Attalla HY, Siddig EE, Mhmoud NA, Musa AM, van de Sande WWJ, Scherrer B, Oyieko P, Egondi TW, Onyango KO, Hata K, Chu WY, Dorlo TPC, Bruggemann RJ, Nyaoke BA, Strub-Wourgaft N, Zijlstra EE. Two dose levels of once-weekly fosravuconazole versus daily itraconazole in combination with surgery in patients with eumycetoma in Sudan: a randomised, double-blind, phase 2, proof-of-concept superiority trial. Lancet Infect Dis. 2024 Nov;24(11):1254-1265. doi: 10.1016/S1473-3099(24)00404-3. Epub 2024 Aug 1. PMID 39098321